CLINICAL TRIAL: NCT06420713
Title: Use of Xenogeneic Bone Graft Associated With Autogenous Bone Graft or Leukocyte-and-Platelet-Rich Fibrin (L-PRF) for Horizontal Bone Augmentation of Alveolar Ridge: A Randomized Controlled Clinical Trial
Brief Title: Horizontal Bone Augmentation of Alveolar Ridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Michel Reis Messora, Associate professor at the department of Oral and Maxillofacial Surgery and Periodontology, School of Dentistry of Ribeirao Preto, University of Sao Paulo-USP, Ribeirao Preto, São Paulo, Brazil, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13102219.0.0000.5419
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Platelet-rich Fibrin; Bone Substitutes; Atrophic Maxilla; Cone-beam Computed Tomography; Bone Regeneration
MeSH Terms: conditions — Atrophic Maxilla | interventions — Population Groups; Dental Implants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autogenous bone graft or Leukocyte-and-Platelet-Rich Fibrin (L-PRF) (Active Comparator)
  Interventions: Procedure: Groups
- Groups (Active Comparator)
  Interventions: Procedure: Horizontal Bone Augmentation of Alveolar Ridge
- Dental Implants (Active Comparator)
  Interventions: Procedure: Dental Implants

INTERVENTIONS:
Procedure: Horizontal Bone Augmentation of Alveolar Ridge — Elevation of the flap in the anterior region of atrophic maxilla to receive particulate autogenous bone mixed with deproteinized bovine bone graft (Group A) or Leukocyte-and-Platelet-Rich Fibrin (L-PRF) mixed with deproteinized bovine bone graft (Group B). In both groups, bone augmentations were covered with a collagen membrane stabilized with pins.
  Arms: Groups
Procedure: Groups — The patients underwent Guided Bone Regeneration (GBR) procedures for the reconstruction of atrophic edentulous alveolar ridges and were divided into two groups according to the proposed treatment:
  Group A - GBR using a mixture of particulate autogenous bone graft and deproteinized bovine bone graft (Bio-Oss® Small; Geistlich AG, Wolhusen, Switzerland).
  Group B - GBR using a mixture of deproteinized bovine bone graft (Bio-Oss® Small) and L-PRF + Liquid Fibrinogen.
  Arms: Autogenous bone graft or Leukocyte-and-Platelet-Rich Fibrin (L-PRF)
Procedure: Dental Implants — After 8 months of GBR healing, dental implants were placed in the grafted regions using guided surgery techniques.
  Cone beam computed tomography (CBCT) scans were performed preoperatively, immediately after the surgical procedure, and after 8 months of follow-up to measure the linear and volumetric changes in the alveolar ridge. At the time of dental implant placement, after an 8-month period following the GBR procedures, bone biopsies were obtained from the grafted area for histological and micro-CT analysis.
  The stability of the implants was assessed using resonance frequency analysis in the immediate postoperative period and at 6 months postoperatively.
  After the 6-month period following dental implant placement, the patients were cleared for implant-supported prosthetic rehabilitation.
  Arms: Dental Implants

SUMMARY:
The objective of this randomized controlled clinical trial was to evaluate the effects of particulate xenogeneic bone grafts associated with autogenous bone graft or Leukocyte-and-Platelet-Rich Fibrin (L-PRF) for horizontal alveolar ridge augmentation. Twenty-eight patients presenting edentulous regions and requiring horizontal bone augmentation prior to dental implant placement were included in this study and randomly divided into two groups according to the proposed guided bone regeneration (GBR) treatment.

Fourteen surgical sites corresponding to Group A received bone regeneration with particulate autogenous bone tissue associated with deproteinized bovine bone graft (Bio-Oss Small®; Geistlich AG, Wolhusen, Switzerland). In Group B, fourteen surgical sites were regenerated with deproteinized bovine bone graft (Bio-Oss Small®) associated with L-PRF. In both groups, the grafted region was protected by a collagen membrane (Bio-Gide® Compressed; Geistlich AG, Wolhusen, Switzerland) fixed to the buccal and palatal bone plates using titanium pins.

Cone-beam computed tomography (CBCT) scans were performed preoperatively, immediately after the GBR surgical procedure, after 8 months of GBR healing, and immediately after dental implant placement to measure linear and volumetric changes in the alveolar ridge. At the time of dental implant placement, after an average period of 8 months following the guided bone regeneration procedures, bone biopsies were taken from the grafted area for histological, histomorphometric, and micro-CT analysis.

After a period of 6 months, the dental implants were reopened to receive implant-supported prosthetic rehabilitation. Implant stability was assessed using resonance frequency analysis at the time of implant placement in the grafted area and after an average of 6 months during the reopening surgical stage. Patient pain perception following bone regeneration procedures was assessed using a visual analog scale. All obtained data were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* a requirement for the placement of one to four dental implants exclusively in the maxilla;
* insufficient horizontal bone remaining for dental implant placement (maximum width of 4mm);
* sufficient vertical bone height for subsequent placement of dental implant(s).

Exclusion Criteria:

* any contraindication for dental implant placement;
* the need for vertical bone augmentation;
* inflammatory or autoimmune disease in the oral cavity;
* use of immunosuppressants, corticosteroids, or bisphosphonates;
* a history of malignancy in the past 5 years;
* smokers;
* patients reporting excessive alcohol consumption;
* decompensated systemic condition;
* uncontrolled periodontal disease;
* insulin-dependent diabetic patients;
* patients with blood-related diseases.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Micro-CT and Histometric analyses | 8 months
  After the period of 8 months from Horizontal Bone Augmentation of Alveolar Ridge, during the dental implant placement by guided surgery, bone samples will be collected at the same location of the implants preparation. The collected bone tissue will be prepared and submitted to Micro-CT and histometric analyses.

SECONDARY OUTCOMES:
Dental Implants ISQ measurement | 6 months
  ISQ will be measured at the moment of implant placement and after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry of Ribeirão Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No